CLINICAL TRIAL: NCT06772298
Title: Study of Oxidized Albumin in Liver Transplant Patients
Acronym: SALT
Status: Not yet recruiting | Type: Observational
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Other Study IDs: K 2024-3904
Record Dates: First submitted 2024-06-03; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-05

CONDITIONS: Liver Failure; Liver Cirrhosis; Liver Transplant Disorder
Keywords: Oxidised albumin; Complement; Coagulation
MeSH Terms: conditions — Liver Failure; Liver Cirrhosis; Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and serum samples will be obtained
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall goal is to describe the oxidation state of albumin before, during and after liver transplantation. This is a pilot observational study in which the oxidative state in 10 patients undergoing liver transplantation will be described. Samples for analysing the oxidation state of albumin, general oxidative damage and anti-oxidant state, the activation of the complement system and factors involved in coagulation will be obtained before transplantation, before and after reperfusion of the portal vein and on postop days 1, 2 and about 30.

ELIGIBILITY:
Inclusion Criteria:

* Patients on waiting list for liver transplantation

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient that are accepted for liver transplantation and put on the waiting list will be included
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Albumin quality | Before transplantation, before and after reperfusion of the portal vein and on postop days 1, 2 and about 30.
  Describe potential qualitative changes in albumin during the liver transplantation procedure. Non-oxidised, single oxidised and double oxidised albumin will be analysed by HPLC.

SECONDARY OUTCOMES:
Effect of clinical factors on albumin quality before transplantation | Before transplantation.
  Explore the impact of different clinical factors on albumin's oxidative state before transplantation. For this a multiple regression model will be used including clinical parameters; sex (male or female), age (years), and MELD (Model for end-stage liver disease).
Effect of clinical factors on albumin quality after transplantation | On postop days 1, 2 and about 30.
  Explore the impact of different clinical factors on albumin's oxidative state after transplantation. For this a multiple regression model will be used including clinical parameters; sex (male or female), age (years), MELD (Model for end-stage liver disease), bleeding during surgery (in liters), time of surgery (hours).
Graft outcome in relation to albumin quality | At days 1, 2 and about 30 days after transplantation
  Explore of the oxidation state of albumin (percentage of albumin that is oxidised) is correlated with graft function (bilirubin levels in mg/L)
Oxidative stress in relation to albumin quality | Before transplantation, before and after reperfusion of the portal vein and on postop days 1, 2 and about 30.
  Explore is the oxidation state of albumin (percentage of albumin oxidised) is related to a general oxidative state measured by TBARS (Thiobarbituric acid reactive substances) measured as MDA (malondialdehydes) in nmol/ml.
Anti-oxidant capacity in relation to albumin quality | Before transplantation, before and after reperfusion of the portal vein and on postop days 1, 2 and about 30.
  Explore is the oxidation state of albumin (percentage of albumin oxidised) is related to the total anti-oxidant capacity measured a the ability of the sample to reduce ferric ions (Fe3+) to ferrous ions (Fe2+) using a phenanthroline substance.
Binding capacity | Before transplantation, before and after reperfusion of the portal vein and on postop days 1, 2 and about 30.
  Explore whether the oxidation state of albumin (percentage of albumin oxidised) is affecting albumin's binding capacity measured by the ability of albumin in the sample to bind cobalt (mg/ml).
Complement system | Before transplantation, before and after reperfusion of the portal vein and on postop days 1, 2 and about 30.
  Explore how the complement system (C3bc in mg/ml) is affected during liver transplantation and how this is related to albumin quality (percentage of albumin oxidised)
Complement system | Before transplantation, before and after reperfusion of the portal vein and on postop days 1, 2 and about 30.
  Explore how the complement system (terminal complement complex in mg/ml) is affected during liver transplantation and how this is related to albumin quality (percentage of albumin oxidised)
Coagulation | Before transplantation, before and after reperfusion of the portal vein and on postop days 1, 2 and about 30.
  Explore how coagulation (Thrombin-antithrombin complex in microgram/ml) is affected during liver transplantation and how this is related to albumin quality (percentage albumin oxidised)

IPD SHARING:
Plan to Share IPD: Undecided
Data might be shared on special request of researchers